CLINICAL TRIAL: NCT01489371
Title: A Phase I Study of Intraperitoneal Egen-001 (IL-12 Plasmid Formulated With PEG-PEI-Cholesterol Lipopolymer) Administered in Combination With Pegylated Liposomal-Doxorubicin (PLD, Doxil (NSC# 712227 or Lipodox (NSC#673089) in Patients With Recurrent or Persistent Epithelial Ovarian, Fallopian Tube or Primary Peritoneal Cancer
Brief Title: EGEN-001 and Pegylated Liposomal Doxorubicin Hydrochloride in Treating Patients With Recurrent or Persistent Ovarian Epithelial Cancer, Fallopian Tube Cancer, or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOG-9928; NCI-2012-00088 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000719230; GOG-9928 (Other: NRG Oncology); GOG-9928 (Other: CTEP); U10CA180868 (NIH); U10CA027469 (NIH); NCT01673477 (obsolete NCT alias)
Record Dates: First submitted 2011-12-08; First posted 2011-12-09 (Estimated); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Ovarian Clear Cell Cystadenocarcinoma; Ovarian Endometrioid Adenocarcinoma; Ovarian Seromucinous Carcinoma; Ovarian Serous Cystadenocarcinoma; Ovarian Undifferentiated Carcinoma; Recurrent Fallopian Tube Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Primary Peritoneal Carcinoma
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — GEN-1; liposomal doxorubicin; Doxorubicin

ARMS (1):
- Treatment (EGEN-001, pegylated liposomal doxorubicin) (Experimental): Patients receive pegylated liposomal doxorubicin hydrochloride IV over 60 minutes on day 1 and EGEN-001 IP over 30-60 minutes on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: PEG-PEI-cholesterol Lipopolymer-encased IL-12 DNA Plasmid Vector GEN-1; Drug: Pegylated Liposomal Doxorubicin Hydrochloride

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: PEG-PEI-cholesterol Lipopolymer-encased IL-12 DNA Plasmid Vector GEN-1 — Given IP
  Other Names: GEN-1; IL-12 Plasmid Formulated With PEG-PEI-Cholesterol Lipopolymer; Nanoparticle-encased IL-12 DNA Plasmid Vector; phIL-12-005
Drug: Pegylated Liposomal Doxorubicin Hydrochloride — Given IV
  Other Names: ATI-0918; Caelyx; DOX-SL; Doxil; Doxilen; Doxorubicin HCl Liposome; doxorubicin hydrochloride liposome; Duomeisu; Evacet; LipoDox; Liposomal Adriamycin; liposomal doxorubicin hydrochloride; Liposomal-Encapsulated Doxorubicin; Pegylated Doxorubicin HCl Liposome; S-Liposomal Doxorubicin; Stealth Liposomal Doxorubicin; TLC D-99

SUMMARY:
This phase I trial studies the side effects and the best dose of giving EGEN-001 together with pegylated liposomal doxorubicin hydrochloride in treating patients with ovarian epithelial, fallopian tube, or primary peritoneal cancer that has returned after a period of improvement or has not responded to treatment. Biological therapies, such as EGEN-001, may stimulate the immune system in different ways and stop tumor cells from growing. Drugs used in chemotherapy, such as pegylated liposomal doxorubicin hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving EGEN-001 together with pegylated liposomal doxorubicin hydrochloride may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum-tolerated dose (MTD) and dose-limiting toxicities (DLTs) of EGEN-001 when administered in combination with pegylated liposomal doxorubicin hydrochloride (PLD; Doxil; Lipodox) every 28 days and the associated DLTs based on adverse events that occur in cycle 1 for this combination in women with recurrent or persistent epithelial ovarian, fallopian tube, or primary peritoneal cancer.

II. To examine the tolerability of the combination at the MTD of EGEN-001 assessed in combination with PLD.

III. To determine recommended phase II dose (RP2D) of EGEN-001 in combination with PLD.

SECONDARY OBJECTIVES:

I. To estimate the objective response rate (complete and partial) in patients with measurable disease.

TERTIARY OBJECTIVES:

I. Determine the levels and time course of interleukin-12 (IL-12), interferon-gamma (IFN-gamma), tumor necrosis factor-alpha (TNF-alpha) and vascular endothelial growth factor (VEGF) following EGEN-001 treatment.

II. Assess the effect of EGEN-001 treatment on the nature of the cellular immune responses by measuring cell-specific ribonucleic acid (RNA) transcripts.

OUTLINE: This is a dose-escalation study of EGEN-001.

Patients receive pegylated liposomal doxorubicin hydrochloride intravenously (IV) over 60 minutes on day 1 and EGEN-001 intraperitoneally (IP) over 30-60 minutes on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up quarterly for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologic diagnosis of epithelial ovarian, fallopian tube, or primary peritoneal carcinoma which is now persistent or recurrent; histologic documentation of the original primary tumor is required via the pathology report
* Patients with the following histologic epithelial cell types are eligible: high-grade serous adenocarcinoma, endometrioid adenocarcinoma, undifferentiated carcinoma, clear cell adenocarcinoma, mixed epithelial carcinoma, or adenocarcinoma not otherwise specified (N.O.S.)
* Patients must have recurrence documented by elevated CA-125 (biochemical recurrence) or clinically evident measurable or non-measurable recurrent disease as defined below:

  * Biochemical recurrence is defined as a CA-125 greater than or equal to two times the upper normal limit; patients whose CA-125 is less than 100 U/mL must undergo a second confirmatory value within a period of not more than 4 weeks; patients with a level greater than or equal to 100 U/mL may be entered without confirmatory measurement; the CA-125 assessment for eligibility must be done at least 4 weeks after paracentesis or other surgical procedures
  * Detectable (non-measurable) disease is defined as symptomatic ascites or pleural effusions, solid and/or cystic abnormalities on radiographic imaging that do not meet RECIST 1.1 definitions for target lesions and/or biopsy-proven recurrence
  * Measurable disease will be defined by RECIST 1.1; measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded); each lesion must be ? 10 mm when measured by computed tomography (CT), magnetic resonance imaging (MRI), or caliper measurement by clinical exam; or ? 20 mm when measured by chest x-ray; lymph nodes must be ? 15 mm in short axis when measured by CT or MRI

    * Patients with measurable disease must have had at least one ?target lesion? to be used to assess response on this protocol as defined by RECIST 1.1; tumors within a previously irradiated field will be designated as ?non-target? lesions unless progression is documented or a biopsy is obtained to confirm persistence at least 90 days following completion of radiation therapy
* Absolute neutrophil count (ANC) >= 1,500/mcl; this ANC cannot have been induced or supported by granulocyte colony-stimulating factors
* Platelets >= 100,000/mcl
* Creatinine =< 1.5 times institutional upper limit of normal (ULN)
* Bilirubin =< 1.5 times ULN
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 3.0 x ULN
* Alkaline phosphatase =< 2.5 x ULN
* Left ventricular ejection fraction (LVEF) greater than or equal to institutional lower limit of normal (LLN) as determined by gated cardiac radionucleotide scan (multi-gated acquisition scan [MUGA]) or echocardiogram
* Neuropathy (sensory and motor) less than or equal to grade 1
* Patients must have recovered from effects of recent surgery, radiotherapy, or chemotherapy
* Patients should be free of active infection requiring parenteral antibiotics
* Any hormonal therapy directed at the malignant tumor must be discontinued at least one week prior to registration; continuation of hormone-replacement therapy is permitted
* Any other prior therapy directed at the malignant tumor, including biological and immunologic agents, must be discontinued at least three weeks prior to registration
* Patients must have had one prior platinum-based chemotherapeutic regimen for management of primary disease containing carboplatin, cisplatin, or another organoplatinum compound; this initial treatment may have included intraperitoneal therapy, consolidation, non-cytotoxic agents, or extended therapy administered after surgical or non-surgical assessment
* Patients are allowed to receive, but are not required to receive, two additional cytotoxic regimens for management of recurrent or persistent disease, with no more than 1 non-platinum, non-taxane regimen
* Prior treatment with pegylated liposomal doxorubicin hydrochloride [Doxil] or other anthracyclines is NOT allowed
* Patients are allowed to receive, but are not required to receive, non-cytotoxic therapy (such as bevacizumab) as part of their primary treatment regimen
* Patients who have received only one prior cytotoxic regimen (platinum-based regimen for management of primary disease), must have a platinum-free interval of less than 12 months, have progressed during platinum-based therapy, or have persistent disease after a platinum-based therapy
* Gynecology Oncology Group (GOG) performance status of 0 or 1
* Patients of childbearing potential must have a negative pregnancy test prior to the study entry and be practicing an effective form of contraception; if applicable, patients must discontinue breastfeeding prior to study entry
* Patients who have met the pre-entry requirements
* Patients must have signed an Institutional Review Board (IRB)-approved informed consent and authorization permitting release of personal health information

Exclusion Criteria:

* Patients who have received prior treatment with EGEN-001
* Patients who have received prior PLD, doxorubicin, or other anthracyclines
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to EGEN-001 or other agents used in this study
* Patients who have received oral or parenteral corticosteroids within 2 weeks of study entry or who have a clinical requirement for ongoing systemic immunosuppressive therapy
* Patients receiving treatment for active autoimmune disease; ?active? refers to any condition currently requiring therapy; examples of autoimmune disease include systemic lupus erythematosus, multiple sclerosis, inflammatory bowel disease and rheumatoid arthritis
* Patients with other invasive malignancies, with the exception of non-melanoma skin cancer and other specific malignancies as noted below are excluded if there is any evidence of other malignancy being present within the last three years; patients are also excluded if their previous cancer treatment contraindicates this protocol therapy
* Patients who have received prior radiotherapy to any portion of the abdominal cavity or pelvis are excluded; prior radiation for localized cancer of the breast, head and neck, or skin is permitted, provided that it was completed more than three years prior to registration, and the patient remains free of recurrent or metastatic disease
* Patients who have received prior chemotherapy for any abdominal or pelvic tumor (other than ovarian, fallopian tube and primary peritoneal) are excluded; patients may have received prior adjuvant chemotherapy for localized breast cancer, provided that it was completed more than three years prior to registration, and that the patient remains free of recurrent or metastatic disease
* Patients with known active hepatitis
* Patients with concurrent severe medical problems unrelated to the malignancy that would significantly limit full compliance with the study or expose the patient to extreme risk or decreased life expectancy
* Patients of childbearing potential, not practicing adequate contraception, patients who are pregnant, or patients who are breastfeeding are not eligible for this trial
* Patients with history or evidence upon physical examination of central nervous system (CNS) disease, including primary brain tumor, seizures not controlled with standard medical therapy, any brain metastases, or history of cerebrovascular accident (CVA, stroke), transient ischemic attack (TIA) or subarachnoid hemorrhage within six months of the first date of treatment on this study
* Uncontrolled hypertension, defined as systolic > 140 mm Hg or diastolic > 90 mm Hg
* Myocardial infarction or unstable angina within 6 months prior to registration
* History of serious ventricular arrhythmia (i.e., ventricular tachycardia or ventricular fibrillation) or cardiac arrhythmias requiring anti-arrhythmic medications (except for atrial fibrillation that is well controlled with anti-arrhythmic medication)
* Corrected QT (QTc) interval >= 450 ms on baseline EKG (electrocardiogram)
* Baseline ejection fraction =< 50% as assessed by echocardiogram or multi gated acquisition scan (MUGA)
* New York Heart Association (NYHA) class II or higher congestive heart failure
* Grade 2 or higher peripheral ischemia (brief [< 24 hrs] episode of ischemia managed non-surgically and without permanent deficit)
* Patients with any condition/anomaly that would interfere with the appropriate placement of the IP catheter for study drug administration including: abdominal surgery within 4 weeks of study entry (for reasons other than IP port placement), intestinal dysfunction, or suspected extensive adhesions from prior history or finding at laparoscopy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-07-09 (Actual); Primary Completion 2014-12-30 (Actual); Study Completion 2018-01-27 (Actual)

PRIMARY OUTCOMES:
First course DLTs | 28 days
The grade of toxicity as assessed by CTCAE v 4.0 | Up to 1 year

SECONDARY OUTCOMES:
Objective tumor response (complete and partial response) | Up to 1 year

OTHER OUTCOMES:
Change in biomarker levels | Baseline to up to 1 year
  Descriptive statistics and graphics will be used to examine the time course of changes.
Change in cellular immune response as measured by cell-specific RNA transcripts | Baseline to up to 1 year
  Descriptive statistics and graphics will be used to examine the time course of changes.

CONTACTS AND LOCATIONS:
Overall Officials: Premal H Thaker, Principal Investigator — NRG Oncology
Locations (7):
- United States (7):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Washington University School of Medicine, St Louis, Missouri
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Case Western Reserve University, Cleveland, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin